CLINICAL TRIAL: NCT02174783
Title: The Safety and Efficacy of Mediterranean Diet and Protein-Sparing Modified Diet on Obesity and Metabolic Syndrome in Liver Transplant Recipients: A Randomized Clinical Trial
Brief Title: Mediterranean Diet and Protein-Sparing Modified Diet for Metabolic Syndrome in Liver Transplant Recipients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTMS-9500
Record Dates: First submitted 2014-06-23; First posted 2014-06-26 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2014-07

CONDITIONS: Liver Transplantation; Metabolic Syndrome X; Obesity
Keywords: Weight Loss; Diet, Mediterranean; Diet, Reducing; protein sparing modified diet
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Weight Loss | interventions — Control Groups; Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (Active Comparator): Standard of care group
  Interventions: Other: Control group
- Mediterranean diet (Experimental): Mediterranean diet for 6 months
  Interventions: Other: Mediterranean diet
- Protein-Sparing Modified Fast (PSMF) (Experimental): PSMF for 6 months
  Interventions: Other: Protein-Sparing Modified Fast (PSMF)

INTERVENTIONS:
Other: Control group — Patient will be provided with basic nutrition educational materials that outline principles of a healthy diet, including: moderation, portion control, increased intakes of fruits, vegetables and whole grains and reduced intakes of saturated fat, salt and sugar. Brief education will be provided by the hepatologist without dietitian referral.
  Arms: Control group
Other: Mediterranean diet — Patient will receive verbal diet instruction from the dietitian or from the hepatologist who has received instruction from the dietitian on following the Mediterranean diet.
  Arms: Mediterranean diet
Other: Protein-Sparing Modified Fast (PSMF) — Patient will be referred to the dietitian for an appointment to discuss the PSMF plan.
  Protein needs of 1.5 grams/kilogram will be calculated based on patient's actual body weight.
  Patient will receive verbal instruction from the dietitian, as well as printed materials for reference at home. Dietitian will provide a list of allowed and prohibited foods as per Cleveland Clinic's PSMF diet standards.
  Arms: Protein-Sparing Modified Fast (PSMF)

SUMMARY:
Many metabolic complications can develop after liver transplant including: diabetes, high blood pressure, obesity, heart attacks and stroke. The goal of this study is to look at the safety and effect of 2 well known and established diet regimens on the people who had a prior liver transplant and investigate whether it helps with the control of these comorbidities.

DETAILED DESCRIPTION:
The Mediterranean diet has been shown to be effective in improving hepatic steatosis, insulin sensitivity, diabetes control and reducing cardiovascular risk in adult patients, but there is no data available for patients who underwent liver transplant. The protein-sparing modified fast (PSMF) diet has been used for years at the Cleveland Clinic to treat adult patients with obesity-related medical problems, but its safety and efficacy has not been established in liver transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

Adult patients > 18 years old who had a successful liver transplant at least 1 year prior to enrollment who also have a BMI>30 with previous failed attempts at weight loss via conventional methods. In addition to one of the following:

1. Triglyceride (TG)>150 mg/dl or specific treatment for this lipid abnormality
2. HDL <40 mg/dl in females and <50 mg/dl in males or specific treatment of this lipid abnormality
3. Systolic BP >130 or diastolic BP >85 mm Hg or treatment for previously diagnosed hypertension
4. Fasting plasma glucose >100 mg/dl or previously diagnosed type 12 diabetes

Exclusion Criteria:

* Significant behavioral issues that would interfere with compliance
* Lack of readiness to change (pre-contemplation, contemplation or preparation stages)
* Previous bariatric surgery
* Pregnant or planning to become pregnant
* History of a documented eating disorder (e.g. bulimia)
* History of kidney stones

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Weight loss | 6 months

SECONDARY OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events | 6 months
  Investigate the safety of the mediterranean diet and PSMF in post liver transplant patients
Change in Hb A1c compared to baseline | 6 months
Change in HDL and LDL compared to baseline | 6 months
Change in triglyceride compared to baseline | 6 months
Change in blood pressure compared to baseline | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: mohammed Eyad Yaseen Alsabbagh, MD, Principal Investigator — The Cleveland Clinic; Naim Alkhouri, MD, Study Director — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States